CLINICAL TRIAL: NCT03109119
Title: Does Sevoflurane Induce Genomic Instability in Patients Undergoing General Anaesthesia?
Brief Title: Does Sevoflurane Cause Genomic Damage
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jubilee Mission Medical College and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 08/16/IEC / JMMC&RI
Record Dates: First submitted 2017-03-20; First posted 2017-04-12 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Anesthesia; Adverse Effect
Keywords: genomic instability; Sevoflurane; General anaesthesia
MeSH Terms: conditions — Genomic Instability | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Intervention Model Description: All children will be randomly allocated into two groups - group S and P. Children in group S will be anaesthetised with sevoflurane, whereas children in group P will be anaesthetised with propofol.
  Peripheral blood samples of 1.5 ml each will be taken immediately after extubation (S-2) , after 48 hours (S-3)and after 120 hours (S-4).A fifth blood sample (S-5) will be taken on the 14th postoperative day.
  These blood samples will be evaluated for genomic instability using Alkaline Comet Assay and micronucleus test by the Genetics Lab of our hospital.
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a double blinded study, where the participants are randomly selected using a computer - generated number and allocated to any one of the two groups. Both the patient and the outcome assessor will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group S (Active Comparator): These patients will be induced and maintained with sevoflurane during anaesthesia.
  Interventions: Drug: Sevoflurane
- Group P (Sham Comparator): These patients will be induced and maintained with propofol during anaesthesia.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — The patients in the group S will be exposed to routine concentrations of sevoflurane during anaesthesia.
  Other Names: sevorane
  Arms: Group S
Drug: Propofol — These patients will be induced with propofol 1.5 mg / kg and maintained with propofol infusion.
  Other Names: fresofol
  Arms: Group P

SUMMARY:
This study aims to find out if sevoflurane causes any cell damage to patients undergoing general anaesthesia. In case of any damage, the reversibility of the damage is also assessed. This is a prospective, comparative study carried out in all children scheduled for surgical repair of cleft lip or palate admitted in the Department of Plastic Surgery under Smile Train organisation ìn our hospital,who satisfy the inclusion and exclusion criteria.

DETAILED DESCRIPTION:
STUDY GOALS AND OBJECTIVES

1. To find out if sevoflurane induces genomic instability in children undergoing cleft lip and palate repair.
2. To assess the magnitude of genomic damage caused by the sevoflurane anaesthesia.
3. To evaluate the reversibility of the induced genomic instability when exposure is discontinued.

STUDY DESIGN Type of study : Prospective Comparative Study Research population : All children scheduled for surgical repair of cleft lip or palate admitted in the Department of Plastic Surgery of our hospital, who satisfy the inclusion and exclusion criteria.

Sample Size : A total of 30 children will be enrolled for the study. METHODOLOGY Children scheduled to undergo surgical repair of cleft lip or palate were enrolled for the study, after addressing the inclusion and exclusion criteria.

A peripheral blood sample of 1.5 ml (S-1) will be taken before the induction of anaesthesia .All children will be randomly allocated into two groups - group S and P.All children will be premedicated with Inj.Glycopyrolate 0.01 mg/kg . Children in group S will be induced with sevoflurane, whereas children in group P will be induced with propofol.All children will be intubated using I / V Vecuronium 0.1 mg / kg .Analgesia will be provided using I / V Fentanyl 1.5 mcg / kg. Depth of anaesthesia will be maintained with sevoflurane in group S and with propofol infusion in group P. The vitals will be monitored as usual intraop and the children will be extubated at the end of the surgery.

Peripheral blood samples of 1.5 ml each will be taken immediately after extubation (S-2) , after 48 hours (S-3)and after 120 hours (S-4).A fifth blood sample (S-5) will be taken on the 14th postoperative day All the blood samples will be evaluated for genomic instability using Alkaline Comet Assay by the Genetics Lab of our hospital.

STATISTICAL ANALYSIS

The findings of this study will be analysed using Chi-square test, Student's t-test, Mann-Whitney U test, mean and standard deviation to yield the final results. The study will be considered statistically significant with a p value of less than 0.05

ELIGIBILITY:
Inclusion Criteria

* Children must have isolated cleft lip or palate.
* The surgery must be a primary repair of cleft lip or palate.
* The minimum duration of the surgery must be 90 minutes.

Exclusion Criteria

* Children who have undergone previous surgery.
* Children who have syndromic cleft lip or palate.
* Children with bleeding disorders.
* Children with known allergy to any of the concerned drugs.

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Genomic instability | It will be assessed at 2 hours after anaesthesia.
  Genomic instability will be assessed using comet assay
Genomic instability | It will be assessed 48 hours after anaesthesia.
  Genomic instability will be assessed using comet assay.

SECONDARY OUTCOMES:
Reversibility of the genomic instability | It will be assessed on fifth day after anaesthesia.
  Assessed using comet assay
Reversibility of genomic instability | It will be assessed on the 14th day after anaesthesia.
  It will be assessed using comet assay.

CONTACTS AND LOCATIONS:
Overall Officials: Vigil Peter, MD, Principal Investigator — Jubilee Mission Medical College and Research Institute, Thrissur, India
Locations (1):
- Jubilee Mission Medical College and Research Institute, Thrissur, Kerala, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Szyfter K, Szulc R, Mikstacki A, Stachecki I, Rydzanicz M, Jaloszynski P. Genotoxicity of inhalation anaesthetics: DNA lesions generated by sevoflurane in vitro and in vivo. J Appl Genet. 2004;45(3):369-74. PMID 15306730
- [Result] Musak L, Smerhovsky Z, Halasova E, Osina O, Letkova L, Vodickova L, Polakova V, Buchancova J, Hemminki K, Vodicka P. Chromosomal damage among medical staff occupationally exposed to volatile anesthetics, antineoplastic drugs, and formaldehyde. Scand J Work Environ Health. 2013 Nov;39(6):618-30. doi: 10.5271/sjweh.3358. Epub 2013 Mar 22. PMID 23525098
- [Result] Fenech M, Holland N, Chang WP, Zeiger E, Bonassi S. The HUman MicroNucleus Project--An international collaborative study on the use of the micronucleus technique for measuring DNA damage in humans. Mutat Res. 1999 Jul 16;428(1-2):271-83. doi: 10.1016/s1383-5742(99)00053-8. PMID 10517999
- [Result] Wiesner G, Schiewe-Langgartner F, Lindner R, Gruber M. Increased formation of sister chromatid exchanges, but not of micronuclei, in anaesthetists exposed to low levels of sevoflurane. Anaesthesia. 2008 Aug;63(8):861-4. doi: 10.1111/j.1365-2044.2008.05498.x. Epub 2008 Jun 6. PMID 18540930
- [Result] Tania K.de Araujo, Roseane L, Flora M.B.B, Nilson C.R, Cristina W.P, Ricardo Manoel da Cruz et al-Genotoxic effects of anaesthetics in OT personnel evaluated by micronuclei tests Journal of Anaesthesia and Clinical Science ISSN 2049-9752,10.7243/2049-9752-2-26,2013
- [Result] Rozgaj R, Kasuba V, Brozovic G, Jazbec A. Genotoxic effects of anaesthetics in operating theatre personnel evaluated by the comet assay and micronucleus test. Int J Hyg Environ Health. 2009 Jan;212(1):11-7. doi: 10.1016/j.ijheh.2007.09.001. Epub 2007 Nov 26. PMID 18023252
- [Result] Alcaraz M, Quesada S, Armero D, Martin-Gil R, Olivares A, Achel GD. Genotoxicity and cytotoxicity of sevoflurane in two human cell lines in vitro with ionizing radiation. Colomb Med (Cali). 2014 Sep 30;45(3):104-9. eCollection 2014 Jul-Sep. PMID 25386035
- [Result] Braz MG, Braz LG, Barbosa BS, Giacobino J, Orosz JE, Salvadori DM, Braz JR. DNA damage in patients who underwent minimally invasive surgery under inhalation or intravenous anesthesia. Mutat Res. 2011 Dec 24;726(2):251-4. doi: 10.1016/j.mrgentox.2011.09.007. Epub 2011 Sep 16. PMID 21944903